CLINICAL TRIAL: NCT00234455
Title: An Evaluation of the Sirolimus-Coated BX VELOCITY Balloon-Expandable Stent in the Treatment of Patients With Bifurcation Lesions.
Brief Title: A Study of the Cypher Sirolimus-Eluting Stent to Treat Bifurcation Lesions.
Acronym: BIFURCATION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll - Medical Affairs Director, Cordis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC01-02
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2008-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): stent in the main branch with balloon angioplasty by a kissing balloon technique in the side branch (stent/PTCA group)
  Interventions: Device: drug eluting-stent
- 2 (Other): stents in both the main and side branches (stent/stent group)
  Interventions: Device: drug-eluting stent

INTERVENTIONS:
Device: drug eluting-stent — PCI
  Other Names: sirolimus-coated Bx VELOCITY Balloon-Expandable Stent
  Arms: 1
Device: drug-eluting stent — PCI
  Other Names: sirolimus-coated Bx VELOCITY Balloon-Expandable Stent
  Arms: 2

SUMMARY:
The objective of this study is to assess the feasibility and safety of the sirolimus-coated Bx VELOCITY Balloon-Expandable Stent in treating patients with true bifurcation lesions.

DETAILED DESCRIPTION:
This is a prospective, randomized study that will be conducted at up to 5 centers in Europe and the US. All patients who meet the eligibility criteria will be treated with the sirolimus-coated Bx VELOCITY Balloon-Expandable Stent and Stent Delivery System (SDS). As a secondary objective, patients will be randomized in a 1:1 ratio to receive one stent in the main branch with balloon angioplasty by a kissing balloon technique in the side branch (stent/PTCA group), or to receive stents in both the main and side branches (stent/stent group). It is anticipated that up to 70% of the patients enrolled in the stent/PTCA group will be considered treatment failures and require a stent in the side branch. These patients will have a sirolimus-coated stent placed in the side branch and will be followed per the protocol, but will be analyzed separately. Therefore, it is anticipated that up to 75 patients will be enrolled in the trial. All patients will have repeat angiography at six months, with clinical follow-up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II) OR has documented silent ischemia;
2. Involves a single treatment of a de novo bifurcation lesion in native coronary arteries of patients with single or multivessel disease; patients with multiple lesions can be included only if other lesions treated during the index procedure are successfully treated prior to the treatment of the bifurcation lesion;
3. Has a true bifurcation lesion defined as stenosis > 50% in both the main branch and the ostium of the side branch;
4. Has a main branch vessel that is <=2.5 mm and <=3.5 mm in diameter by on-line QCA proximal to the bifurcation;
5. Has a side branch vessel that is <=2.5 mm and <=3.5 mm in diameter by on-line QCA.

Exclusion Criteria:

1. Patient has experienced a Q-wave or non-Q-wave myocardial infarction with documented elevation of CK levels > 2 times normal or CK-MB levels > 3 times normal within the preceding 24 hours and/or the CK and CK-MB enzymes remain above normal at the time of treatment;
2. Has unstable angina classified as Braunwald A I-III, or III B or C, or is having a peri infarction;
3. Has a bifurcation lesion in a non protected left main;
4. Has an ejection fraction <=35%;
5. There is presence of thrombus in the bifurcation lesion;
6. Has a totally occluded vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2001-06; Primary Completion 2002-10 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
percent residual diameter stenosis (%DS) in the stented branch as measured by quantitative coronary angiography (QCA) | 6-months post-procedure

SECONDARY OUTCOMES:
device success defined as achievement of a final residual diameter stenosis of < 50% (by QCA), using the assigned device/treatment only | anytime during the course of the study
procedure success defined as achievement of a final diameter stenosis of < 50% (by QCA) using any percutaneous method, without the occurrence of death, myocardial infarction (MI), or repeat revascularization of the target lesion during the hospital stay | anytime during the course of the study
target vessel failure (TVF), defined as a composite of cardiac death, MI, or target vessel revascularization | 6, 12, 18, and 24 months post-procedure
lumen and obstruction volume by intravascular ultrasound (IVUS) | 6-month post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Colombo, MD, Principal Investigator — Centre Cuore Columbus
Locations (1):
- Centre Cuore Columbus, Milan, Italy